CLINICAL TRIAL: NCT02743104
Title: Ketamine vs Propofol for Sedation During Pediatric Bronchoscopy
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol being reconsidered
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KP-001
Record Dates: First submitted 2016-04-10; First posted 2016-04-19 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2016-04

CONDITIONS: Paediatric Flexible Bronchoscopy
MeSH Terms: interventions — Ketamine; Propofol; Midazolam; Atropine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine for procedural sedation (Active Comparator): All patients will be sedated according to a written protocol which includes intravenous administration of midazolam and atropine. In addition, local anesthesia will be performed using lidocaine 1% sprayed once just above the vocal cords, and again at the level of the carina. Lidocaine doses are limited to a maximum total dose of 5mg/kg.
  This study group will be exposed to ketamine as the main drug for sedation, as an initial bolus of 1-2 mg/kg initially and then titrated by additional doses of 1mg/kg per dose.
  Interventions: Drug: Ketamine; Drug: midazolam and atropine; Drug: Lidocaine
- Propofol for procedural sedation (Active Comparator): All patients will be sedated according to a written protocol which includes intravenous administration of midazolam and atropine. In addition, local anesthesia will be performed using lidocaine 1% sprayed once just above the vocal cords, and again at the level of the carina. Lidocaine doses are limited to a maximum total dose of 5mg/kg.
  This study group will be exposed to propofol as the main drug for sedation, as an initial bolus of 1-2 mg/kg initially and then titrated by additional doses of 1mg/kg per dose.
  Interventions: Drug: Propofol; Drug: midazolam and atropine; Drug: Lidocaine

INTERVENTIONS:
Drug: Ketamine
  Other Names: Ketalar
  Arms: Ketamine for procedural sedation
Drug: Propofol
  Other Names: Diprivan
  Arms: Propofol for procedural sedation
Drug: midazolam and atropine
Drug: Lidocaine

SUMMARY:
The purpose of this study is to determine whether ketamine or propofol, drugs used for procedural sedation during paediatric bronchoscopy, results in higher operator satisfaction and better side effect profile.

DETAILED DESCRIPTION:
Pediatric bronchoscopy requires moderate to deep sedation in order to maintain patient comfort and safety, while optimizing the working environment for the physician performing the procedure. There is a paucity of pediatric research in the field of pediatric flexible bronchoscopy and data are often extrapolated from adult studies.

Propofol is often used as the sedation drug for this procedure due to its rapid sedative effect and favorable emergence profile. Propofol's major limitation is its tendency to cause apneas, which can occur in a relatively narrow therapeutic window. Apnea risk decreases with the patient's age and administering physician's familiarity and experience with the drug.

Ketamine is a drug often used for pediatric procedural sedation. Its pharmacologic safety profile is very wide, allowing a wide spectrum of dosing with a significantly reduced risk of apnea when compared to propofol. Known adverse effects of the drug include its emergence profile which may be accompanied by hallucinations, bronchorrhea and laryngospasm. Hallucinations may be prevented by using benzodiazepines concurrently and are possibly more pronounced in teenaged children compared to infants, although post-sedation irritability in the latter group might be an expression of this. Bronchorrhea, while usually not of significant concern during procedural sedation, has the potential to play a more noteworthy role during bronchoscopy. Significant airway secretions can create a difficult working environment for the pulmonologist performing the procedure. Patient safety may also be affected, as increased airway secretions reduce visibility in pediatric airways that are narrow to begin with and further compromised by placement of the bronchoscope. Potentially, this might also impact on the child's air flow and gas exchange. Laryngospasm during the procedure potentially hinders passage of the scope beyond the vocal cords and might extend the duration of the procedure.

In the investigators' center, propofol has most often been the sedative drug of choice for bronchoscopy. Yet, ketamine has been used at times due to its safety profile and the administering physicians level of comfort with each drug.

Aim:

To compare operator satisfaction and adverse effects in children presenting for flexible bronchoscopy using ketamine versus propofol as the primary sedative agent.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing flexible bronchoscopy

Exclusion Criteria:

* Failure to acquire parental consent
* Bronchoscopies performed outside of the bronchoscopy suite
* Bronchoscopies performed under general anesthesia with a protected airway
* Bronchoscopies performed by personnel outside of the study group
* Known allergies to either of the sedation drugs used

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Overall Pulmonologist's satisfaction level (VAS) | 2 years
  Assessed via visual analog scale

SECONDARY OUTCOMES:
Amount of airway secretions | 2 years
  Assessed via visual analog scale
Cough score | 2 years
  Assessed via visual analog scale

IPD SHARING:
Plan to Share IPD: Yes
Group data will be published. No individual data will be made available.

REFERENCES:
- [Background] Hwang J, Jeon Y, Park HP, Lim YJ, Oh YS. Comparison of alfetanil and ketamine in combination with propofol for patient-controlled sedation during fiberoptic bronchoscopy. Acta Anaesthesiol Scand. 2005 Oct;49(9):1334-8. doi: 10.1111/j.1399-6576.2005.00842.x. PMID 16146472
- [Background] Dal T, Sazak H, Tunc M, Sahin S, Yilmaz A. A comparison of ketamine-midazolam and ketamine-propofol combinations used for sedation in the endobronchial ultrasound-guided transbronchial needle aspiration: a prospective, single-blind, randomized study. J Thorac Dis. 2014 Jun;6(6):742-51. doi: 10.3978/j.issn.2072-1439.2014.04.10. PMID 24976998
- [Background] Wahidi MM, Jain P, Jantz M, Lee P, Mackensen GB, Barbour SY, Lamb C, Silvestri GA. American College of Chest Physicians consensus statement on the use of topical anesthesia, analgesia, and sedation during flexible bronchoscopy in adult patients. Chest. 2011 Nov;140(5):1342-1350. doi: 10.1378/chest.10-3361. PMID 22045879
- [Background] Stolz D, Chhajed PN, Leuppi J, Pflimlin E, Tamm M. Nebulized lidocaine for flexible bronchoscopy: a randomized, double-blind, placebo-controlled trial. Chest. 2005 Sep;128(3):1756-60. doi: 10.1378/chest.128.3.1756. PMID 16162784